CLINICAL TRIAL: NCT07369999
Title: Effects of Butylphthalide Enhanced With Tenecteplase on Neurological Function in Mild Disabling Acute Ischemic Stroke -A Prospective, Multicenter, Randomized, Double-blind, Active-controlled Trial
Brief Title: Effects of Butylphthalide Enhanced With Tenecteplase on Neurological Function in Mild Disabling Acute Ischemic Stroke
Acronym: BENEFIT-2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202512130
Record Dates: First submitted 2026-01-08; First posted 2026-01-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Mild Disabling Acute Ischemic Stroke
Keywords: Mild Disabling Acute Ischemic Stroke; Butylphthalide; Tenecteplase
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination Group (Experimental)
  Interventions: Drug: Combination Group
- Control Group (Placebo Comparator)
  Interventions: Drug: Control Group

INTERVENTIONS:
Drug: Combination Group — Combination Group: TNK 0.25 mg/kg (maximum 25 mg) administered as a single intravenous infusion. Immediately after that, NBP 100 ml (25 mg) is initiated as an intravenous infusion, twice daily (bid), for 7 consecutive days. If the hospitalization duration is less than 7 days, oral NBP soft capsules (0.2 g, three times daily [tid]) will be started on the day of discharge, and continued until Day 14.
  Arms: Combination Group
Drug: Control Group — Control Group: TNK 0.25 mg/kg (maximum 25 mg) administered as a single intravenous infusion. Immediately after that, a 100 ml intravenous infusion of NBP placebo (visually identical to NBP) is initiated twice daily (bid) for 7 consecutive days. If the hospitalization duration is less than 7 days, oral NBP placebo soft capsules (visually identical, 0.2 g, three times daily [tid]) will be started on the day of discharge and continued until Day 14.
  Arms: Control Group

SUMMARY:
Abstract Background Intravenous thrombolysis is the cornerstone of early treatment for acute ischemic stroke (AIS), but some still have a poor prognosis, especially in patients with mild disabling stroke. Tenecteplase (TNK), a novel thrombolytic agent with favorable pharmacokinetic profiles, and butylphthalide (NBP), a multi-targeted neuroprotective drug, have shown promising efficacy in separate clinical applications. However, evidence for their combined use in mild disabling AIS is lacking.

Aim To determine whether TNK combined with NBP can improve functional outcomes compared with TNK monotherapy in patients with mild disabling AIS who receive thrombolysis within 4.5 hours of onset.

Design BENEFIT-2 is a prospective, multicenter, randomized, double-blind, active-controlled trial. Eligible patients are randomized 1:1 to receive either TNK plus NBP (combination group) or TNK plus placebo (control group) via stratified block randomization. The combination group receives sequential NBP sodium chloride injection (25mg/100ml, twice daily for 7 days) and oral NBP soft capsules (0.2g, three times daily) until day 14; the control group receives matching placebos.

Eligibility criteria include age 18-80 years, onset time ≤4.5 hours, NIHSS score 2-5 with disabling manifestations (hemianopia, aphasia, or limb weakness), and pre-stroke modified Rankin Scale (mRS) score ≤1.

Study outcomes The primary outcome is the proportion of patients with mRS score 0-1 at 90±7 days. Secondary outcomes include changes in NIHSS score, recurrence of ischemic stroke, composite vascular events, quality of life (assessed by EQ-5D scale), and ischemic penumbra salvage rate. Safety outcomes include symptomatic intracranial hemorrhage (sICH), vascular death, all-cause death, and adverse events within 90 days.

Discussion BENEFIT-2 is the first large-scale randomized trial to evaluate the synergistic effect of "vascular recanalization + neuroprotection" in mild disabling AIS. By combining TNK and NBP, this study aims to fill the evidence gap and provide a new therapeutic option to improve functional recovery in this specific population.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-80 years, regardless of gender.
* 2. Clinically diagnosed with acute ischemic stroke and meets the criteria for tenecteplase intravenous thrombolysis.
* 3. Onset of the current stroke within 4.5 hours.
* 4. Clinical diagnosis of minor ischemic stroke with a NIHSS score of 2-5, accompanied by persistent unilateral limb weakness or speech symptoms, defined as a score ≥1 on either the language item or any one limb item of the NIHSS
* 5. Pre-stroke mRS score ≤1.
* 6. The subject or their legal representative is able and willing to sign the informed consent form.

Exclusion Criteria:

* 1. History of intracranial hemorrhage.
* 2. Patients who have received or plan to undergo mechanical thrombectomy.
* 3. History of major head trauma or stroke within the past 3 months.
* 4. Known severe liver/kidney dysfunction or patients receiving dialysis (severe liver dysfunction: ALT/AST >3 times the upper limit of normal; severe kidney dysfunction: serum creatinine >3.0 mg/dl [265.2 μmol/L] or GFR <30 ml/min/1.73 m²).
* 5. Systolic blood pressure <90 mmHg or >220 mmHg.
* 6. Patients with bradycardia (heart rate <60 beats/min) or sick sinus syndrome.
* 7. History of drug/food allergy or known allergy to the components of the study drugs.
* 8. Patients treated with drugs containing butylphthalide after stroke onset.
* 9. History of congenital/acquired hemorrhagic diseases, coagulation factor deficiency, or thrombocytopenic diseases.
* 10. Pregnant or lactating subjects or subjects planning to become pregnant within 90 days.
* 11. Subjects with severe mental disorders or dementia who cannot cooperate with informed consent and follow-up.
* 12. Subjects with concurrent malignant tumors or severe systemic diseases, with an expected survival of <90 days.
* 13. Patients who have participated in other clinical interventional studies within 30 days prior to randomization, or who are currently participating in other clinical interventional studies;
* 14. Patients who are unable to complete follow-up visits as scheduled;
* 15. Any other reasons that, in the investigator's opinion, render the patient unsuitable for participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1062 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Modified Rankin Scale score 0-1 (scores 0 = fully asymptomatic to 6 = death) | From enrollment to the end of treatment at 90 days

SECONDARY OUTCOMES:
proportion of patients with Modified Rankin Scale score 0-2 (scores 0 = fully asymptomatic to 6 = death) | From enrollment to the end of treatment at 90 days
Proportion of patients with National Institutes of Health Stroke Scale score improvement ≥2 points at 90±7 days compared with baseline. (0-42, higher scores indicate more severe neurological impairment) | at 90±7 days compared with baseline.
Changes in National Institutes of Health Stroke Scale score from baseline to 6±1 days and 90±7 days. (0-42 points,higher scores indicate more severe neurological impairment) | From enrollment to 6±1 days and 90±7 days
Incidence of early neurological deterioration (NIHSS score increase ≥4 points) at 24±2 hours and 6±1 days. | From enrollment to 24±2 hours and 6±1 days.
Recurrence rate of ischemic stroke | From enrollment to 90±7 days.
Proportion of composite vascular events (stroke recurrence, myocardial infarction, vascular death) | From enrollment to90±7 days.
Ischemic penumbra salvage rate (change in DWI/PWI mismatch volume from baseline to 6±1 days). | from baseline to 6±1 days
Quality of life assessed by the EQ-5D scale (utility score and visual analog scale) | From enrollment to90±7 days.
Stratified composite endpoint: mRS score 0-1 or NIHSS score improvement ≥2 points | From enrollment to 90±7 days.

OTHER OUTCOMES:
Incidence of serious adverse events within 90 days (Primary safety outcome) | From enrollment to 90 days
  Primary safety outcome: Incidence of serious adverse events within 90 days (defined as events leading to death, life-threatening conditions, hospitalization/prolonged hospitalization, persistent disability, or congenital anomalies).
Symptomatic intracranial hemorrhage at 24±2 hours and 6±1 days; | From enrollment to 24±2 hours and 6±1 days;
Vascular death at 90±7 days; | From enrollment to 90±7 days
All-cause death at 90±7 days | From enrollment to 90±7 days

IPD SHARING:
Plan to Share IPD: No